CLINICAL TRIAL: NCT02115217
Title: Effect of Kinesiotaping on Ankle Stability in a Population of Elite Basketball Players
Brief Title: Effect of Kinesiotaping on Ankle Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Romande de Readaptation (Network)
Collaborators: University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CliniqueRR-02
Record Dates: First submitted 2014-03-14; First posted 2014-04-15 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2015-07

CONDITIONS: Sprain and Strain of Ankle
Keywords: Kinestiotaping; Basketball players; Effect of kinesiotaping; on postural stability
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Leukotape K, basketball training (Experimental): Use of Leukotape K to ensure stability of the ankle in basketball players
  Interventions: Device: Leukotape K
- Sham, basketball training (Placebo Comparator): Use of sham tape
  Interventions: Device: Sham kinesiotape

INTERVENTIONS:
Device: Leukotape K — All interventions will be performed by a qualified physiotherapist in a standardized manner. Tape will be extended to the recommended length (120%) and applied along the outer side of the leg, along the path of the peroneal muscle. Starting in the middle of the foot arch, the tape ends 1 cm below tibial head.
  Other Names: Leukotape K, Johnson & Johnson
  Arms: Leukotape K, basketball training
Device: Sham kinesiotape — KT put with no effects
  Arms: Sham, basketball training

SUMMARY:
Ankles sprains are the most popular injuries in basketball players. They are traumatic injuries, which happen most of the time in specific situations, like landing on another player's foot, or during changes of direction.

Neuromuscular exercises are very important to improve ankle stability and reduce risks of sprains. However various external support such as ankles braces and rigid tape, are also used in order to prevent injury.

The kinesiotape (KT) is a new but broadly used method in the world of athletes. Created by KenzoKase, in 1980, this kind of tape has a tremendous success with athletes and is today commonly used during practices and/or competitions. The main property of this tape is its elasticity, which is supposed to improve proprioception and, thus ankle stability, but these aspects have not been investigated yet.

DETAILED DESCRIPTION:
Aim: Compare the effects of a kinesiotape (KT) with a sham treatment (KT put with no effects) and a control condition (absence of tape) in basketball players from the Swiss national league through balance tests on an unstable surface.

Hypotheses: A KT positioned on the lateral side of the leg improves ankle stability in basketball players while balancing on an unstable surface.

Method: 30 subjects will be recruited from different basketball teams affiliated to the Swiss national league. They will have to perform some postural stability tests on both unstable ("Delos") and stable surfaces ("Single Les Stance", "Star Excursion Balance Test", "Cross Over Hop Test for Distance") under three different conditions. The three condition will be as followed : with a KT positioned on the lateral side of the leg, with a sham tape or without tape. The three sessions will be spaced in time (7 days of wash out). The order of the three interventions (KT, Sham tape, no tape) will be randomized (cross over) to avoid the bias of learning processes. Neither the subjects nor the examiner will be aware of the "tape condition" (double blind); a physiotherapist will be in charge of positioning the tape according to the tested condition.

The sequence of the tests will be the same for all subjects and breaks are scheduled to avoid the effect of the fatigue. An anamnesis of all subjects will be done in order to evaluate history of injuries. At the end of each session, a visual analogical scale will be completed by the athlete to obtain a personal feeling of stability . The subject will be also asked to determine which condition was tested.

Expected results: the application of a KT on the lateral side of the leg improves postural stability on instable surfaces in elite basketball players.

Field's importance: the application of KT may reduce the risk of ankle sprains and the recurrence of sprains in a population of athletes at risk.

ELIGIBILITY:
Inclusion Criteria:

* active elite basketball players

Exclusion Criteria:

* no history of ankle sprain in the last 6 weeks
* no history of any other lower limbs lesion in the last 6 weeks

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of kinesiotaping on postural stability | For each subject outcome will be assessed in the 3 weeks following the beginning of the study.
  To assess postural stability, the following parameters will be measured:
  Autonomy:
  This measure represents the time the subject can stay on the mobile board without the use of his hand to maintain equilibrium.
  Mean axis spacing:
  This measure will be performed using an accelerometer localized on the sternum of the subjects. This device will allow us to calculate displacement of the chest (degrees of inclination).
  Mean error of the board:
  This parameter represents numerically the inclination of the board during the test. It allows to estimate the stability of the subjects' ankle (unit=degrees). The larger this value is the lower the stability will be.
  An estimation of total equilibrium between each subject will be assessed using the two parameters listed here above (mean axis spacing + mean error of the board) following recommendation of the manufacturer.

SECONDARY OUTCOMES:
EVA scale to evaluate the sensation of postural stability | Assessment will be performed within 3 weeks after the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Yan Eggel, MD, Principal Investigator — Clinique Romande de Readaptation; Lia Volpe, Student, Principal Investigator — Institut des Sciences du Sport de l'Université de Lausanne; Olivier Dériaz, Md, PhD, Study Director — Institut de Recherche en Readaptation; Jérôme Barral, PhD, Study Director — Institut des Sciences du Sport de l'Université de Lausanne
Locations (1):
- Clinique Romande de Réadaptation, Sion, Valais, Switzerland